CLINICAL TRIAL: NCT00432471
Title: Evaluation of Optical Imaging for Margin Delineation of Non-Melanoma Skin Cancers
Brief Title: Optical Imaging of Skin Cancers for Margin Delineation of Non-Melanoma Skin Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0493; 1R21DE016485-01 (NIH); NCI-2015-01901 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Skin Cancer
Keywords: Skin Cancer; Non-Melanoma Skin Cancer; Optical Imaging; Multispectral Digital Microscope System; MDM
MeSH Terms: conditions — Skin Neoplasms | interventions — Optical Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Optical Imaging (Experimental): Imaging using the multispectral digital microscope (MDM), a system that shines different colors of light on the skin and takes pictures of fluorescence and reflectance on the skin area.
  Interventions: Procedure: Optical Imaging

INTERVENTIONS:
Procedure: Optical Imaging — Imaging using the multispectral digital microscope (MDM), a system that shines different colors of light on the skin and takes pictures of fluorescence and reflectance on the skin area.

SUMMARY:
The goal of this clinical research study is to evaluate an experimental imaging technology, the multispectral digital microscope (MDM), which may help doctors see how far skin cancer extends (widens out) on an area of skin. Researchers want to learn if this new technology can help doctors identify the exact areas involved in precancerous or cancerous changes in the skin.

DETAILED DESCRIPTION:
All tissue and cells are made of tiny particles that give off small amounts of light. This light is called fluorescence. Researchers have learned that cancerous cells and normal cells give off different amounts and different types of fluorescence. Cancerous cells and normal cells also reflect (bounce back) light differently. Researchers want to better understand if light fluorescence and reflectance (a measure of the ability of a material to reflect sunlight) from the skin can be used to tell which cells may be cancerous.

Researchers have developed the MDM system in order to better understand how cancer changes the light fluorescence and reflectance in skin. The MDM system shines different colors of light on the skin and takes pictures of fluorescence and reflectance on the skin area through a microscope. The pictures will then be studied to better understand the differences in fluorescence and reflectance in abnormal and normal cells.

If you agree to take part in this study, an area of your skin will first be examined under standard white light. A researcher will then use the MDM imaging instrument to take pictures of abnormal-looking and normal skin areas. The researcher will mark 2-4 areas of your skin with a marker. During your surgery, you will have a small sample from a normal-looking area collected and 1 or 2 samples collected, from abnormal-looking areas of the skin. Each sample from abnormal-looking tissue will be about 3-4 millimeters wide (about the size of a small pencil eraser).

After the skin lesion has been removed, but before it is needed for review by the pathologist or surgeon, the removed tissue will be examined using the MDM imaging instrument and standard white light. The edges of the removed lesion will then be examined with another type of microscope, a confocal microscope, which allows researchers to see the very small cells in the tissue. The exact location that was imaged with this microscope will be marked on the tissue, and the findings will be recorded. The tissue will then be checked by the pathologist according to standard procedures.

You will not be told of any of the experimental findings. Information about the diagnosis will be available to your treating doctor.

Your name and any personal identifying information (such as your name, social security number, or medical record number) will be coded to protect your privacy.

This is an investigational study. Up to 55 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be undergoing surgery to remove a region of skin suspected of containing non-melanoma skin cancer will be eligible to participate in this study. The proposed resection should be equal or greater than 1 cm in diameter.
2. In addition, patients undergoing induction chemotherapy or biologic therapy prior to surgical resection are also eligible.
3. Patients must sign an informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

1. Patients with non-melanoma skin cancer lesion at eyelid, or in case that the lesion extends to superior or inferior eyelid, this area will not be imaged.
2. Persons who are medically unfit to undergo resection of skin lesions.
3. Persons under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-01-30 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Evaluate use of fluorescence and reflectance imaging, and confocal microscopy for non-invasive detection of skin tumor margins in head and neck region | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org